CLINICAL TRIAL: NCT02875509
Title: Wound Infammatory Cells After Cardiac Surgery and the Patients´Survival. A Sixteen Years Follow-up Study
Brief Title: Wound Inflammatory Cells After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Turku University
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Sternotomy Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
One hundred patients, aged from 41 to 78 years, underwent open heart surgery in the years 1998-1999 and were studied by using the Cellstick device for harvesting wound inflammatory cells during the first 24 hours after surgery. The results of the differential count were computerized by using artificial neural network for obtaining wound inflammatory cell node (WICN). The patients were followed up for sixteen years or to the death. WICN values were compared with the patients´ survival.

ELIGIBILITY:
Inclusion Criteria:

* Elective operations

Exclusion Criteria:

* Urgency operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergone open heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 1998-03; Primary Completion 1999-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
death | 16 years

CONTACTS AND LOCATIONS:
Overall Officials: Timo JA Savunen, MD, Principal Investigator — Turku University Hospital

IPD SHARING:
Plan to Share IPD: No